CLINICAL TRIAL: NCT02419287
Title: Pilot Study of Crizotinib in Relapsed ALK+ Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRU1
Record Dates: First submitted 2015-04-03; First posted 2015-04-17 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Anaplastic Large Cell Lymphoma, ALK-Positive
Keywords: ALK; crizotinib
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- crizotinib (Experimental): 250mg BID
  Interventions: Drug: crizotinib

INTERVENTIONS:
Drug: crizotinib

SUMMARY:
The purpose of this study is to determine the response and the duration of it in patients affected by ALK+ lymphoma that are resistant or refractory to standard cytotoxic treatment that will be treated with crizotinib.

DETAILED DESCRIPTION:
Study Rationale

Crizotinib is a selective ATP-competitive small-molecule inhibitor of the c-Met/HGFR and ALK receptor tyrosine kinases and their oncogenic variants (eg. c-Met/HGFR mutations or NPM-ALK fusion protein). Consistent with this mechanism of action, Crizotinib inhibited phosphorylation of c-Met/HGFR and NPM-ALK and their kinase target dependent functions in tumour cells both in vitro and in vivo. This compound will be clinically evaluated in oncology indications in which c-Met/HGFR or NPM-ALK are dysregulated including, but not limited to renal, lung, gastric, brain, prostate, head, and neck cancers, multiple myeloma, and selected lymphomas. Crizotinib demonstrated preclinical antitumour activity, including marked cytoreduction, in several tumour models that expressed activated c-Met/HGFR or NPM-ALK, supporting the rationale for study in clinical trials. Collective PK/PD modelling and efficacy data demonstrated that:

1. near complete inhibition (free plasma IC90) of c-Met/HGFR activity during the entire dosing interval was necessary to achieve robust antitumour effect, as it was demonstrated several years ago for imatinib;
2. the target efficacious free plasma concentration range was determined to be 8.1 to 12.8 nM (3.7 to 5.8 ng/mL). The projected efficacious dose in humans is estimated to be 70 to 100 mg once daily.

Additional safety and efficacy data presented at the 2010 ASCO meeting (Tan et al., Bang et al.) confirmed these data: plasma concentrations exceeding efficacious levels were obtained in patients receiving at least 100 mg/day of crizotinib; in addition objective tumour regressions were observed in >50% of 82 advanced lung cancer patients whose tumours were positive for the EML4/ALK fusion. Therefore the treatment of ALK+ lymphomas with crizotinib represents a rational attempt at treating a human cancer through the inactivation of its oncogenic mechanism.

When administered to 11 patients affected by relapsed resistant ALK+ lymphomas, crizotinib obtained an Overall Response Rate (ORR) of 10/11 (91%) which included 9 Complete Responses (CR, 82%) and 1 Partial Response. Disease status at the latest follow-up (June 2013) is as follows: 4 CR (months 17+, 26+, 31+, 36+) and 3 deaths due to progression; 1 patient in CR after crizotinib who received alloBMT and 2 patients (treated post alloBMT) are still in CR but they stopped crizotinib; 1 patient is in CR under brentuximab. Progression Free Survival (PSF) and Overall Survival rates at 3 years are 63.6% and 72.7%. Crizotinib exerted a potent antitumor activity in advanced ALK+ lymphoma and produced durable responses in this population of heavily pre-treated patients. In addition this study demonstrated that PCR-based detection of the NPM-ALK fusion in the peripheral blood may be an effective method to monitor disease response and progression.

Although crizotinib shows activity, relapses occur typically within 5 months after starting treatment and were supported by mutations like I1171N.

Objectives Primary Define the objective response rates (ORR) and duration of it in subjects with ALK+ lymphomas resistant or refractory to standard cytotoxic treatment, according to RECIST 1.1 criteria.

Secondary

* Define progression free survival (PFS) and overall survival (OS) in ALK+ lymphoma patients treated with crizotinib, that are resistant or refractory to standard cytotoxic treatment. Determine the toxicity profile of crizotinib in ALK+ lymphoma patients resistant or refractory to standard cytotoxic treatment.
* Determine the Quality of Life (QoL) in this population of patients using the the EORTC - C30 Quality of Life questionnaire.
* Study the molecular mechanism of resistance to crizotinib.

Study design This is a phase II study open to 12 eligible patients with anaplastic large cell lymphoma with a confirmed ALK rearrangement. Enrollment will start in February 2015 and it will last 24 months.

All patients must have been pretreated with at least one line of standard cytotoxic chemotherapy and they must have demonstrated progression (regardless of initial response) on the last treatment.

Subject selection Before any clinical procedure, patients will sign the Informed Consent. Every patients included in this protocols will have to respect all inclusion/exclusion criteria.

Study procedure The study begins with a screening period to assess eligibility, up to and including 28 days prior to the first dose of crizotinib. The treatment period begins on Day 1 of Cycle 1. Assessments of tumor response will be performed after 1 month, 2 months (only Q-RT-PCR for NPM/ALK), 3 months and then every 12 weeks, starting from the first day of treatment with crizotinib. After 1 year of treatment, assessments will be collected every six months. From the beginning of the third year, assessments will be performed yearly till the end of the study. Clinical, laboratory assessments, Quantitative Real-Time PCR (Q-RT-PCR) and tumor imaging will be performed as described in Appendix 1.

Treatment will continue until patient experiences unacceptable toxicity or progressive disease (PD), starts a new anti-cancer therapy or dies.

When the patient discontinues from study treatment an EOT visit must be performed within 7 days of the last dose of crizotinib. Patients will be contacted for the safety with a follow-up 30 days after their last dose of crizotinib.

During the follow up phase, patients will be contacted once a year to obtain information pertaining to survival status until death, loss to follow-up, withdrawal of consent to survival follow-up, or the end of the study. Patients do not need to visit the clinic during the survival follow-up.

Study Treatment Patients will receive crizotinib at the dose of 250 mg BID administered orally. Crizotinib will be taken at approximately the same time each day.

In case of toxicity, it is possible to proceed to a dose reduction or a temporary interruption of crizotinib according with the attached table (Appendix 2).

No dose escalation is scheduled. The metabolism of crizotinib is predominantly mediated by the CYP3A isozymes in human liver microsomes and hepatocytes. Co-administration with drugs that are CYP3A inhibitors and inducers may change plasma concentration of crizotinib in humans. Concomitant use of potent CYP3A inhibitors or inducers are not allowed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Informed Consent approved by Local Ethical Committee before any protocol-specific screening procedures.
2. ALK+ Non-Hodgkin lymphoma diagnosed by IHC or FISH.
3. Refractory disease or relapse after at least one prior chemotherapy regimen (typically a minimum of 6 cycles of CHOP); presence of measurable disease by physical examination, CT or CT-PET scan.
4. Any prior chemotherapy or major surgeries must have been completed at least 14 days prior to initiation of study medication. This could not be respected if there is clear evidence of disease progression, manifested as growing pain attributable to the tumour, fever, growing tumour lesions, increasing LDH values.
5. Able to take oral therapy.
6. Female or male, 18 years of age or older.
7. ECOG performance status 0-3.
8. Adequate organ function as defined by the following criteria:

   * Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN) or AST and ALT ≤ 5 x ULN if liver function abnormalities are due to underlying malignancy
   * Total serum bilirubin 1.5 x ULN (except patients with documented Gilbert's syndrome
   * Creatinine ≤ 1.5 x ULN.
9. Adequate bone marrow function:

   * Absolute neutrophil count (ANC) ≥ 1000/µL
   * Platelets ≥ 50.000/µL
   * Hemoglobin ≥ 9.0 g/dL The hematological values will not be considered in case of bone marrow involvement.
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
11. Female and male patients who are of childbearing potential must agree to use an effective form of contraception with their partners throughout participation in this study.

Exclusion Criteria:

1. Current treatment on another therapeutic clinical trial.
2. Prior therapy specifically directed against ALK.
3. Major surgery within 14 days prior first dose of crizotinib.
4. History of uncontrolled cardiac disease including: myocardial infarct, uncontrolled angina or hypertension, clinically significant ventricular arrhythmia, unexplained syncope.
5. Pregnancy or breastfeeding.
6. Use of drugs or foods that are known potent CYP3A4 inhibitors, including but not limited to amprenavir, atazanavir, clarithromycin, delavirdine, diltiazem, erythromycin, indinavir, itraconazole, ketoconazole, miconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin, verapamil, voriconazole, and grapefruit or grapefruit juice.
7. Use of drugs that are known potent CYP3A4 inducers, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, rifapentine, tipranavir, ritonavir, and St. John's wort.
8. Use of drugs that are CYP3A4 substrates with narrow therapeutic indices, including but not limited aripiprazole, ergotamine, halofantrine, pimozide, triazolam, astemizole*, cisapride*, and terfenadine* (* withdrawn from U.S. market).
9. Prior malignancy other than basal cell carcinoma.
10. Other severe acute or chronic medical or psychiatric conditions, or laboratory abnormalities that would impart, in the judgment of the investigator and/or sponsor, excess risk associated with study participation or study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
objective response rates (ORR) in subjects with ALK+ lymphomas resistant or refractory to standard cytotoxic treatment, according to RECIST 1.1 criteria. | the entire duration of the study (5 years)
Duration ORR | the entire duration of the study (5 years)

SECONDARY OUTCOMES:
Progression free survival (PFS) in ALK+ lymphoma patients treated with crizotinib, that are resistant or refractory to standard cytotoxic treatment. | the entire duration of the study (5 years)
Number of patients with adverse events after crizotinib treatment | the entire duration of the study (5 years)
Quality of Life (QoL) in this population of patients using the the EORTC - C30 Quality of Life questionnaire | the entire duration of the study (5 years)
Overall survival (OS) in ALK+ lymphoma patients treated with crizotinib | the entire duration of the study (5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gambacorti Passerini, MD, Principal Investigator — University of Milano Bicocca
Locations (1):
- ASST-Monza, Monza, Italy/MB, Italy

REFERENCES:
- [Result] Rindone G, Aroldi A, Bossi E, Verga L, Zambrotta G, Tarantino S, Piazza R, Mussolin L, Chiarle R, Gambacorti-Passerini C. A monocentric analysis of the long-term safety and efficacy of crizotinib in relapsed/refractory ALK+ lymphomas. Blood Adv. 2023 Feb 14;7(3):314-316. doi: 10.1182/bloodadvances.2022007538. No abstract available. PMID 35914224